CLINICAL TRIAL: NCT04354064
Title: Circulating Tumor DNA (ctDNA) for Early Treatment Response Assessment of Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Roche Sequencing Solutions (Industry); The Foundation for Barnes-Jewish Hospital (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); Radiological Society of North America (Other); Skandalaris (Unknown); The V Foundation for Cancer Research (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201903142
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer; Prostate Cancer; Head and Neck Cancer; Esophageal Cancer; Genitourinary Cancer; Sarcoma; Breast Cancer; Colon Cancer; Gastrointestinal Cancer; Solid Tumor Cancer; Lung Cancer; Skin Cancer; Melanoma
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms; Urogenital Neoplasms; Sarcoma; Breast Neoplasms; Colonic Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms; Skin Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * Blood and/or urine from healthy volunteers under this study
  * The remaining samples (tissue, blood, drain fluid, urine, plasma) will be collected under various repository and banking studies at Washington University School of Medicine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Donor Samples: * Donation of blood and/or urine samples as often as bi-monthly and as many as 24 times in total
  * These samples will be used to generate reference data to compare patient data to and/or to correct stereotypic noise.
- Samples from Repository and Banking Studies: * Healthy prostate and/or blood and/or urine samples from Genitourinary Repository
  * Tissue, blood, and/or drain fluid samples from Head and Neck Banking studies
  * Tissue and/or blood samples from Esophageal Repository
  * Tissue and/or blood samples from Genitourinary Repository
  * Tissue and/or plasma from Sarcoma Tissue Bank
  * Tissue and/or plasma from Breast Cancer Bank
  * Tissue, plasma, and/or urine from GI Tissue and Blood Bank
  * Tissue, blood, and/or urine from Solid Tumor Bank
  * Tissue, blood, and/or urine from Lung Cancer Bank
  * Tissue and/or blood from Skin Cancer Bank
  * Tissue and/or blood from Pediatric Neurosurgery Tissue Bank

SUMMARY:
Earlier detection of disease recurrence will enable greater treatment options and has strong potential to improve patient outcomes. This project is translational and has the potential to lead to future translational research opportunities, including interventional trials in which therapeutic escalation is offered at the early circulating tumor DNA (ctDNA) molecular residual disease (MRD) detection timepoint. Ultimately, the integration of ctDNA into the clinical workflow has the potential to enhance cancer diagnosis, treatment, surveillance, and prognosis, and guide clinical decision-making in this era of personalized precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Eligible healthy donors will be at least 18 years of age.

Exclusion Criteria:

* Healthy donors younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * This study will access data and specimens from patients who consented to specimen banks (approximately 3262 patients) There is a waiver of consent for this study regarding patient data banked under the tissue banks.
  * Healthy donors will be consented prior to sample acquisition (approximately 100 patients)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from progression | Through completion of study (estimated to be 6.5 years)
  -Defined as RECIST 1.1 based radiographic or clinical progression, with non-progressors censored at last radiographic follow-up

SECONDARY OUTCOMES:
Event-free survival | Through completion of study (estimated to be 6.5 years)
  -Defined as post-treatment ctDNA detection or RECIST 1.1 based radiographic progression
Disease-specific survival | Through completion of study (estimated to be 6.5 years)
  -Defined as death from cancer
Overall survival | Through completion of study (estimated to be 6.5 years)
  -Defined as death from any cause
Pathologic complete response rate | Through completion of study (estimated to be 6.5 years)
Locoregional failure | Through completion of study (estimated to be 6.5 years)
  -Defined as clinical or radiographic progression within the localized tumor/treatment area or regional lymph nodes
Distant-metastasis-free survival | Through completion of study (estimated to be 6.5 years)
  -Defined as clinical or radiographic progression outside the localized tumor/treatment area and regional lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Reimers, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be available for sharing with other researchers.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu